CLINICAL TRIAL: NCT04001023
Title: Overcoming Chemoresistance in Advanced Ovarian Cancer Via Targeting Hypoxia
Acronym: OVANOX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15867
Record Dates: First submitted 2019-01-11; First posted 2019-06-27 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Carcinoma; Hypoxia
Keywords: advanced ovarian cancer; EF5-PET/CT; hypoxia
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms; Hypoxia | interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PDS (Experimental): 18F-EF5 PET/CT and 18F-FDG PET/CT scan prior to primary cytoreductive surgery and targeted sample collection during primary cytoreductive surgery
  Interventions: Device: Imaging with 18F-EF5 PET/CT
- IDS (Experimental): 18F-EF5 PET/CT and 18F-FDG PET/CT scans prior to diagnostic laparoscopy and after neoadjuvant chemotherapy before interval cytoreductive surgery .
  Targeted sample collection during diagnostic laparoscopy and interval cytoreductive surgery
  Interventions: Device: Imaging with 18F-EF5 PET/CT

INTERVENTIONS:
Device: Imaging with 18F-EF5 PET/CT — Both 18F-FDG PET/CT and 18F-EF5 PET/CT imaging are performed in 1) preoperative work-up to clarify the disease distribution, 2) before IDS to evaluate treatment response to NACT (IDS arm); targeted samples from hypoxic and non-hypoxic tumors are collected during surgery
  Other Names: Collection of targeted samples during surgery

SUMMARY:
The goal of this non-randomized prospective study is to use 18F-EF5-PET/CT imaging to identify and locate intraabdominal hypoxic ovarian cancer lesions. With targeted surgical sampling, precisely obtain hypoxic and potentially chemoresistant cancer tissue for our analyses and identify key molecular differences between hypoxic and non-hypoxic tumors within the same patient.

A portion of advanced stage EOC are inoperable at diagnosis and can be treated with neoadjuvant chemotherapy (NACT) before surgery. This approach offers a unique opportunity to study how hypoxic tumor areas respond to treatment.

DETAILED DESCRIPTION:
MORE SPECIFIC AIMS

1. To validate the feasibility of PET-tracer EF5 in EOC imaging.

   * Quantify the amount and exact locations of hypoxic tumors in EOC patients using herein developed protocol and tracers (18F-EF5 and 18F-FDG) in diagnostic and neoadjuvant settings.
   * Measure the non-cancer related EF5 accumulation spots and establish the potential pitfalls in abdominal EF5 imaging
   * Establish a method to verify hypoxic locations with 18F-EF5-PET/CT information during the operation.
   * Develop and validate a model that predicts chemotherapy response based on functional imaging information.
2. To reveal hypoxia related alterations in collected tissue samples (i.e. altered DNA damage repair, altered mitochondrial respiratory functioning, overexpression of hypoxia response elements etc)

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed advanced epithelial ovarian, primary peritoneal or fallopian tube cancer.
* age 18-79 years
* informed concent

Exclusion Criteria:

* previous cancer
* pregnancy or nursing

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2017-03-09 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
18F-EF5 maximum standardized uptake values (SUVmax) | 2-3 years
  Tumor and musculus gluteus maximus SUVmax ratio ≥1.5 is considered to refer to hypoxia

SECONDARY OUTCOMES:
Correlation between the uptake of 18F-EF5 isotope in PET/CT and immunohistochemical profile of tumor tissue | 2-3 years
Disease-free survival | 5 years
Overall survival | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University hospital, Turku, Finland